CLINICAL TRIAL: NCT04764136
Title: Reliability and Validity of a New Device Measuring Spinal Rotation on the Transverse Plane
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Georgios Krekoukias, Post doctoral researcher, University of Athens
Other Study IDs: 18221
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Scoliometer (scolioscope) — Individuals with scoliosis will participate in this study. The device will be used to determine spinal rotation on the transverse plane. Repeated measures will be taken.

SUMMARY:
The purpose of this research is to investigate the reliability and validity of a new device similar to a scoliometer. The intended name of the device will be Scolioscope

DETAILED DESCRIPTION:
Οne cohort of participants will be used and the reliability of the equipment will be used to test/retest the repeatability of the measurements

The validity will be measured against a gold standard for measuring angles

ELIGIBILITY:
Inclusion Criteria: lumbar and thoracic scoliosis -

Exclusion Criteria: recent spinal surgery, cancer, spinal fixation

-

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anyone with thoracic and/or lumbar scoliosis
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Reliability | 2021-2022
  Reliability of device on repeated measures both intra and inter observer
Validity | 2021-2022
  Validity of device will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Soultanis, MD, Study Chair — Attikon University Hospital, Athens, Greece; GEORGIOS KREKOUKIAS, PT, PhD, Principal Investigator — PT, PhD
Locations (1):
- Motus Liberi Physiotherapy Centre, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided